CLINICAL TRIAL: NCT02652689
Title: Transthoracic Parametric Doppler Assessment of Lung Doppler Signals in Acute Pulmonary Embolism
Brief Title: Diagnosis of Pulmonary Embolism by Doppler Signals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOP023
Record Dates: First submitted 2016-01-05; First posted 2016-01-12 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; pulmonary disease; Lung Doppler signals
MeSH Terms: conditions — Pulmonary Embolism; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic ultrasound (Experimental): Recording Doppler ultrasound signals noninvasively from the right chest wall
  Interventions: Radiation: Diagnostic ultrasound radiation

INTERVENTIONS:
Radiation: Diagnostic ultrasound radiation — Recording Doppler ultrasound signals from the right chest wall

SUMMARY:
The LDS may contain information of significant diagnostic and physiological value regarding the pulmonary parenchyma and vasculature, as well as the cardio- vascular system in general. In pilot clinical studies of patients with acute decompensated heart failure (ADHF) as well as patients with Pulmonary Hypertension, LDS signals patterns unique to these conditions were identified. We believe that these newly discovered ultrasound signals might provide a non-invasive radiation-free means to diagnose and monitor patients with Pulmonary Embolism.

The purpose of this study is to assess the utility of noninvasive assessment of lung Doppler signals performed via transthoracic parametric Doppler. The objective of the study is to evaluate the lung Doppler signals (LDS) in patients diagnosed with acute PE, in order to determine the potential assessment value of this non-invasive method in this potentially life threatening condition.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute PE on CTA

Exclusion Criteria:

* Pregnant women
* Inability to consent
* Patients with severe chest wall deformity
* Previously diagnosed PE
* Pneumonia
* Pulmonary edema
* Pneumothorax
* Severe COPD (gold class III, IV)
* Hemodynamically unstable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Identify lack of Lung Doppler signals in specific lung sections that were diagnosed obstructed by CT | 30min
  The obstructed sections will be compared with healthy lung sections

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gaitini, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided